CLINICAL TRIAL: NCT06027723
Title: Effects of Acute Nicotine Administration on Motivational Mechanisms
Brief Title: Nicotine and Pavlovian Bias
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, John Robert Monterosso, Assoc Prof Psychology, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UP-23-00575
Record Dates: First submitted 2023-08-16; First posted 2023-09-07 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Nicotine Vaping; Nicotine Dependence
Keywords: Nicotine
MeSH Terms: conditions — Vaping; Tobacco Use Disorder | interventions — Nicotine

STUDY DESIGN:
Intervention Model Description: The participant will be randomized to receive either the regular vape with nicotine or the placebo nicotine vape first and will complete a standardized vaping session with the assigned vape. Each participant will receive both vape conditions, one at each laboratory visit. Moreover, they will not know the order of administration.
  After completing the vaping session, participants will be instructed on how to complete a version of the Go/No-Go task. They will see geometrical shapes on the screen, each of which will signal a particular trial type: go-win-win-reward, no-go-to-win-reward, go-to-avoid-losing, or no-go-to-avoid-losing. Participants will be explicitly instructed that the color of the cue edge will correspond to a specific trial: green will represent a "win reward" condition and red will represent an "avoid losing" condition.
Who Masked: Participant, Investigator
Masking Description: Vapes will be color coded and data recorded by color. Correspondence between color and condition will be unblinded at completion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nicotine (Experimental): Participants will follow a standard vape protocol designed to deliver the approximate nicotine typically consumed from 1 cigarette (1.25 mg)
  Interventions: Drug: Nicotine
- Placebo (Placebo Comparator): Participants will follow a standard vape protocol that is equal inhalation to that used in the nicotine condition.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Nicotine — Nicotine delivered through a vape
  Arms: Nicotine
Other: Placebo — Placebo nicotine-free vaping liquid delivered through a vape
  Arms: Placebo

SUMMARY:
Nicotine remains a major cause of health problems in the US and around the world. Insight into the behavioral changes induced by nicotine use may help advance the understanding of the mechanisms underlying the maintenance of nicotine addiction and thus the important factors involved in the quitting process. Pavlovian bias is a phenomenon that includes an approach tendency toward rewarding cues and an action withdrawal tendency in response to punishments. This phenomenon may be particularly relevant to nicotine users. The current study will use an experimental, within-subjects, repeated-measured design to investigate whether acute nicotine administration influences individual Pavlovian bias in nicotine users. By recruiting participants from the University of Southern California (USC) community and contacting participants of previous nicotine-related studies of the Addiction and Self-Control Laboratory at USC, the investigators will enroll forty adult nicotine users in the study. Participants will come to the lab twice after a 10-hour nicotine fast. At each lab visit, participants will undergo a vaping session prior to completing the study tasks. The content of the e-liquid in the vape will vary by nicotine content: the vape will either contain nicotine or not. Subsequent to vaping, participants will complete a version of the Go/No-Go task which will measure their individual levels of Pavlovian bias. The investigators will compare performance on the task across the two conditions within each participant: on- and off- nicotine, after controlling for nicotine withdrawal and nicotine tolerance. Based on past research on nicotine, the researchers anticipate that acute nicotine administration will be associated with higher levels of Pavlovian bias, compared to the off-nicotine condition. Specifically, two patterns are expected to arise: a higher likelihood of making a go-response in the "win reward" condition and a higher likelihood of making a no-go response in the "avoid losing" condition, regardless of whether it is a "go" or "no-go" trial. Participants will also complete a measure of their working memory capacity. The investigators will conduct exploratory analyses for the relationship between different nicotine conditions and working memory capacity.

DETAILED DESCRIPTION:
Nicotine remains a major cause of health problems in the US and around the world. Insight into the behavioral changes induced by nicotine use may help advance the understanding of the mechanisms underlying the maintenance of nicotine addiction and thus the important factors involved in the quitting process. Pavlovian bias is a phenomenon that includes an approach tendency toward rewarding cues and a tendency to withdraw from action in response to punishments. This phenomenon may be particularly relevant in the context of addiction and impulsive behavior patterns. The current project proposes to examine Pavlovian bias in the context of nicotine use. Specifically, the study aims to explore whether acute nicotine administration affects Pavlovian bias among nicotine users.

Previous studies suggest that Pavlovian bias is a universal phenomenon, but that some individuals are better at overcoming it. Nicotine has been shown to make individuals more sensitive to cues that predict loss and reward. Therefore, it is hypothesized that nicotine will increase individuals' existing Pavlovian bias levels.

Moreover, understanding whether nicotine indeed does impact Pavlovian bias may provide insight into ways in which this bias affects nicotine addiction. For example, nicotine use commonly coexists with other substance use behaviors. If nicotine acutely increases Pavlovian bias, this mechanism could partially explain the general increase of impulsive behaviors among nicotine users.

Purpose/Objectives/Aims/Research Questions The primary aim is to explore the effects of acute nicotine administration on Pavlovian bias. After showing eligibility to take part in the study, participants will come to the lab twice, each after a (self-reported) 10-hour abstinence from nicotine. After completing assessments of nicotine withdrawal and nicotine tolerance, participants will complete a standardized vaping bout, either with a vape with nicotine ("on-nicotine") or a denicotinized one ("off-nicotine"). Although the exact dose of inhaled nicotine depends on the particular puff topography of participants, the standardized vape protocol is designed to deliver approximately 2mg of nicotine. Participants will be encouraged to stop if they feel they are on the verge of having any negative nicotine response (e.g., feeling some nausea). Pavlovian bias will then be assessed via performance on a version of the Go/No-Go task. Specifically, the investigators will record participants' response accuracy on each of the four trials: go-to-win-reward, no-go-to-win-reward, go-to-avoid-losing, and no-go-to-avoid-losing. Finally, participants will complete a measure of their working memory capacity. The researchers will compare performance on the task across the two conditions within each participant: on- and off- nicotine, after controlling for nicotine withdrawal and nicotine tolerance. The investigators will also conduct exploratory analyses to determine whether participants' working memory capacity is affected by the different nicotine conditions.

Aim: Examine the effects of acute nicotine administration on Pavlovian bias. The investigators will explore the effects of acute nicotine on "go-bias" and "no-go bias." They anticipate that some level of Pavlovian bias will be observed across both sessions, on- and off- nicotine. Two patterns are expected to arise: a higher likelihood of making a go-response in the "win reward" condition and a higher likelihood of making a no-go response in the "avoid losing" condition, regardless of whether it is a "go" or "no-go" trial. However, after acute nicotine administration, participants will exhibit higher levels of Pavlovian bias, compared to the off-nicotine condition.

Understanding whether nicotine indeed does impact Pavlovian bias may provide insight into ways in which this bias affects nicotine addiction.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years old
* Current nicotine user (at least monthly use over the past 3 months)
* Reported willingness to abstain from all nicotine for at least 10 hours prior to the two lab visits
* English Language Competency

Exclusion Criteria:

- Currently pregnant, planning to become pregnant, or breastfeeding

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Levels of Pavlovian Bias measured through a version of the Go/No-Go task | 0 hours after using the vaping device (right after)
  Participants will complete a version of the Go/No-Go task, which allows to measure individual levels of Pavlovian bias. Pavlovian bias is a phenomenon that includes an approach tendency toward rewarding cues and a tendency to withdraw from action in response to punishments. In the task, participants choose a response (go or no-go) for various visual cues which have specific response-dependent outcomes.The Go/No-Go task design allows to collect participants' task accuracy scores (task accuracy will signify how many correct cue-dependent responses participants make).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Will post data on Open Science Framework
Supporting Information: Study Protocol, SAP, ICF
Time Frame: after publication or 1 year after completion (whichever comes first)
Access Criteria: open
URL: https://osf.io/

REFERENCES:
- [Background] Algermissen J, Swart JC, Scheeringa R, Cools R, den Ouden HEM. Striatal BOLD and Midfrontal Theta Power Express Motivation for Action. Cereb Cortex. 2022 Jul 12;32(14):2924-2942. doi: 10.1093/cercor/bhab391. PMID 34849626
- [Background] Guitart-Masip M, Chowdhury R, Sharot T, Dayan P, Duzel E, Dolan RJ. Action controls dopaminergic enhancement of reward representations. Proc Natl Acad Sci U S A. 2012 May 8;109(19):7511-6. doi: 10.1073/pnas.1202229109. Epub 2012 Apr 23. PMID 22529363
- [Background] Scholz V, Hook RW, Kandroodi MR, Algermissen J, Ioannidis K, Christmas D, Valle S, Robbins TW, Grant JE, Chamberlain SR, den Ouden HEM. Cortical dopamine reduces the impact of motivational biases governing automated behaviour. Neuropsychopharmacology. 2022 Jul;47(8):1503-1512. doi: 10.1038/s41386-022-01291-8. Epub 2022 Mar 8. PMID 35260787
- [Background] Swart JC, Frobose MI, Cook JL, Geurts DE, Frank MJ, Cools R, den Ouden HE. Catecholaminergic challenge uncovers distinct Pavlovian and instrumental mechanisms of motivated (in)action. Elife. 2017 May 15;6:e22169. doi: 10.7554/eLife.22169. PMID 28504638